CLINICAL TRIAL: NCT06058910
Title: Bilistick Point-of-care System 2.0 Bilirubin Validation Utilizing Blood Samples Collected in Pediatric Patients
Brief Title: Bilistick Point-of-care System 2.0 Bilirubin Validation
Status: Completed | Type: Observational
Sponsor: Kettering Health Network (Other)
Collaborators: Bilimetrix s.r.l. (Other)
Responsible Party: Principal Investigator, Jonathan Toot, Principal Investigator, Kettering Health Network
Other Study IDs: KHN-2023-109
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Screening; Kernicterus; Newborn Jaundice; Point-of-Care Testing
MeSH Terms: conditions — Kernicterus; Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn: This study will include newborn pediatric patients under 2-weeks of age who are necessary to conduct this study and are representative of the target population for use with this device.
  Interventions: Diagnostic Test: Bilistick System 2.0 point-of-care testing device

INTERVENTIONS:
Diagnostic Test: Bilistick System 2.0 point-of-care testing device — The routine standard-of-care blood sample collection involves a 0.5 milliliter whole blood draw by the heel stick method for bilirubin assessments under current reference clinical methodology for total bilirubin. An additional 0.035 milliliter of whole blood will be collected for measurement in the point-of-care Bilistick System 2.0 (Bilistick point-of-care testing device). The resulting Bilistick System 2.0 data (i.e., total bilirubin) will be recorded, but will not be entered into the patients' electronic medical records or used for any diagnostic or medical decision purposes.
  Other Names: Bilistick point-of-care testing device

SUMMARY:
This is a validation study involving the Bilistick System 2.0 point-of-care bilirubin measuring device. The validation will be conducted by comparing bilirubin measurements utilizing the standard-of-care blood sample collected for both a diagnostic reference device and Bilistick System 2.0 point-of-care device. Whole blood samples collected from male or female newborns (<2-weeks of age) born at a Kettering Health Network facility to obtain a total of 80 valid comparison pairs between the reference device and the Bilistick System 2.0 point-of-care device with current laboratory standards.

DETAILED DESCRIPTION:
The investigators propose a prospective diagnostic validation study comparing total bilirubin values measured under the reference clinical methodology to the point-of-care Bilistick System 2.0 testing device. During the routine standard-of-care whole blood sample collection (0.5 milliliters whole blood draw) for bilirubin assessments under reference clinical methodology, an additional 0.035 milliliters of whole blood will be collected (not to exceed more than 2 sample collections per week) for measurement in the point-of-care Bilistick System 2.0. The resulting Bilistick System 2.0 data will be recorded, but will not be entered in the patients' electronic medical records or used for any diagnostic or medical decision purposes.

Whole blood samples collected from male or female newborns (<2-weeks of age) born at a Kettering Health Network facility to obtain a total of 80 valid comparison pairs between the reference device and the Bilistick System 2.0 point-of-care device will be included on study.

Consent forms will be Institutional Review Board (IRB)-approved and the parent or legal guardian of the participant will be asked to read the document. The investigator or delegated study staff will explain the research study to the parent or legal guardian of the participant and answer any questions that may arise. A verbal explanation will be provided to allow for the comprehension of the purposes, procedures, and potential risks of the study and rights of the research participant. The parent or legal guardian of the participant will be informed that participation is voluntary, they can withdraw at any time. Sufficient opportunity will be provided to carefully review the written consent form and ask questions prior to signing. The parent or legal guardian of the participant will sign the informed consent document prior to any procedures being done specifically for the study.

Since this study uses blood collected during an existing standard of care blood collection (i.e., there will be NO separate research-specific heel stick) this study poses no additional risk and parental permission will be required by only one parent.

ELIGIBILITY:
Inclusion Criteria:

* Participant is <2-weeks of age
* Participant is inpatient hospital status
* Participant undergoing routine blood sample collection for total serum bilirubin

Exclusion Criteria:

* Parent or legal guardian of participant is Non-English speaking or reading
* Parent or legal guardian of participant unable to give informed consent/parental permission

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will include newborn pediatric patients under 2-weeks of age who are necessary to conduct this study and are representative of the target population for use with this device.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Bilistick Total Bilirubin | birth through 2-weeks of age
  Measurement of total bilirubin (milligram/deciliter) using the Bilistick 2.0 point-of-care system
Reference Clinical Total Bilirubin | birth through 2-weeks of age
  Measurement of total bilirubin (milligram/deciliter) using standard laboratory clinical instrument sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Toot, MD, Principal Investigator — Kettering Health
Locations (1):
- Kettering Health Main Campus, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No